CLINICAL TRIAL: NCT07310862
Title: Gamma Sensory Stimulation (GSS) for Improving Fatigue in People With Multiple Sclerosis
Brief Title: Virtual Reality - Gamma Sensory Stimulation for Improving Fatigue in People With Multiple Sclerosis
Acronym: VR-GSS
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Clarity Health Technologies, Inc (Industry)
Collaborators: Parc de Salut Mar (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CHT0002
Record Dates: First submitted 2025-12-16; First posted 2025-12-30 (Actual); Last update posted 2026-02-03 (Actual); Status verified 2026-01

CONDITIONS: Multiple Sclerosis
Keywords: Fatigue; MS fatigue; Cognitive Fatigue; Mental Fatigue; GSS; Gamma Sensory Stimulation; VR-GSS; Virtual Reality; MFIS; Neuromodulation; 40Hz
MeSH Terms: conditions — Multiple Sclerosis; Fatigue; Mental Fatigue

STUDY DESIGN:
Intervention Model Description: Participants with multiple sclerosis and significant fatigue are randomized (1:1) to receive either active Gamma Sensory Stimulation (GSS) or sham stimulation for 4 weeks in a parallel-group design.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Participants, care providers, treating investigators, and outcome assessors are blinded to treatment allocation. Active and sham stimulation are delivered through identical virtual reality content and session procedures, and no perceptual cues are provided that would allow participants or study staff to distinguish between treatment conditions. Device configuration (active or sham mode) is preset by unblinded technical personnel who are not involved in participant interaction, clinical assessments, or data analysis.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Gamma Sensory Stimulation (Active Comparator): Participants receive Gamma Sensory Stimulation delivered through a virtual reality (VR) headset and headphones. Stimulation sessions last 30 minutes and are delivered four times per week for four weeks within standardized, engaging VR environments.
  Interventions: Device: Virtual Reality Gamma Sensory Stimulation
- Sham Sensory Stimulation (Sham Comparator): Participants receive sham sensory stimulation delivered through a virtual reality (VR) headset and headphones. Sessions last 30 minutes and are delivered four times per week for four weeks within the same VR environments used in the active intervention.
  Interventions: Device: Virtual Reality Sham Sensory Stimulation

INTERVENTIONS:
Device: Virtual Reality Gamma Sensory Stimulation — Participants receive 30 minutes of Gamma Sensory Stimulation delivered through a virtual reality (VR) headset and headphones. Visual and auditory stimulation parameters are configured to deliver rhythmic sensory stimulation intended to engage gamma-band neural activity. Sessions occur four times per week for four weeks and are embedded within standardized VR environments.
  Other Names: 40 Hz sensory stimulation; 40 Hz audiovisual stimulation; Gamma flickers; 40Hz flickers; VR-GSS
  Arms: Gamma Sensory Stimulation
Device: Virtual Reality Sham Sensory Stimulation — Participants receive 30 minutes of sham sensory stimulation delivered through a virtual reality (VR) headset and headphones. The sham intervention uses identical VR environments, session duration, and procedures as the active intervention, providing an equivalent participant experience without delivering therapeutic stimulation. Sessions occur four times per week for four weeks.
  Other Names: sham sensory stimulation; sham VR-GSS
  Arms: Sham Sensory Stimulation

SUMMARY:
This is a double-blind, parallel, randomized, sham-controlled pilot study evaluating the safety, feasibility, and efficacy of Gamma Sensory Stimulation (GSS) delivered via a Virtual Reality (VR) headset in individuals with Multiple Sclerosis (MS) who experience moderate to severe fatigue. Participants will be randomized (1:1) to 4 weeks of active GSS or sham stimulation, followed by a 4-week post-treatment follow-up. The primary objective is to determine whether GSS reduces fatigue, measured by the Modified Fatigue Impact Scale (MFIS). Secondary outcomes include additional fatigue scales, cognitive performance, quality-of-life measures, tolerability and safety.

DETAILED DESCRIPTION:
Gamma Sensory Stimulation (GSS) is a non-invasive audiovisual neuromodulation method that delivers synchronized 40 Hz stimulation to engage gamma-band neural oscillations. Gamma-frequency activity is implicated in cognitive processing and large-scale network coordination, which may be disrupted in people with Multiple Sclerosis (MS), particularly in those experiencing fatigue. Prior research suggests that gamma-frequency entrainment may modulate neural network activity and support functional outcomes.

This single-center, double-blind, randomized, sham-controlled pilot study investigates whether 4 weeks of GSS delivered through an immersive Virtual Reality (VR) system can reduce fatigue in individuals with MS. Participants with moderate to severe fatigue will be randomized in a 1:1 ratio to receive either active GSS or sham stimulation embedded in matched VR content. The intervention consists of 16 in-lab stimulation sessions delivered over 4 weeks (4 sessions per week). Each session includes 30 minutes of active stimulation within a standardized VR experience.

The primary endpoint is the change in Modified Fatigue Impact Scale (MFIS) total score from baseline to End of Treatment (Week 4). Secondary endpoints include changes from baseline to End of Treatment (Week 4) and follow-up (Week 8) in additional validated fatigue measures (Fatigue Severity Scale, Visual Analogue Scale for Mental Fatigue, PROMIS Fatigue), cognitive performance assessed by the Symbol Digit Modalities Test (SDMT), quality-of-life measures (Neuro-QoL Fatigue), and the rate of change in Daily Fatigue Severity (DFS) across the treatment period. Exploratory outcomes include MFIS subscale scores, variability in daily fatigue ratings, embedded cognitive task performance during stimulation, and treatment acceptability.

Safety and tolerability will be assessed through monitoring of adverse events, session attendance, and retention. Electroencephalography (EEG) will be collected at baseline and at End of Treatment (Week 4) for exploratory characterization of neural responses to gamma-frequency stimulation.

This pilot investigation aims to generate preliminary safety, feasibility, and efficacy data to inform future multisite studies evaluating VR-based GSS as a potential at-home therapeutic approach for MS-related fatigue.

ELIGIBILITY:
Inclusion Criteria:

1. Be between 18 to 65 years of age (inclusive) on the day of signing informed consent.
2. Have MS (McDonald criteria 2017) with Modified Fatigue Impact Scale (MFIS) score greater than 33 OR fatigue greater than 4 (out of 7) on the Fatigue Severity Scale (FSS).
3. Sufficient hearing and vision.
4. Any type of disease modifying therapy is allowed and should be stable in the last 3 months.
5. Not having received corticosteroids the previous month.
6. Each subject must sign the informed consent form, in accordance with local requirements, after the scope and nature of the investigation have been explained to the subject, and before Screening assessments.
7. Based on the investigator's judgment, the subject should:

   1. Be able to speak, read, and understand the language of the trial staff and the informed consent form;
   2. Possess the ability to respond verbally to questions, follow instructions, and complete study assessments;
   3. Be able to adhere to the stimulation protocol and visit schedules.
8. Women of child-bearing potential* must have a negative urine pregnancy test before the inclusion in the study and agree to use highly effective contraceptive methods during the study. Highly effective contraceptive methods will include intrauterine device, implant, patch or pill, bilateral tubal occlusion, vasectomized partner and sexual abstinence.

Exclusion Criteria:

1. Any condition or therapy impairing trial participation and assessments.
2. The presence of a relapse or use of IV steroids for any reason 3 months prior to screening visit.
3. Severe systemic diseases or history of cancer or hereditary familiar cancer.
4. Clinically relevant concomitant disease: cardiac, gastrointestinal, hepatic, pulmonary, neurological, renal or other major disease.
5. A history of seizure or epilepsy.
6. Pregnant or breastfeeding women.
7. Drug or alcohol abuse.
8. Patients with active systemic bacterial, viral or fungal infections, or known to have uncontrolled AIDS or to be HIV-positive but not receiving anti-retroviral therapy based on medical history or available clinical information at screening.
9. Dementia or severe psychiatric, cognitive or behavioral problems or other comorbidity that may interfere with the compliance to the protocol.
10. Any other clinically relevant medical or surgical condition, which, in the opinion of the investigator, would put the subject at risk by participating in the study.
11. Participation in other experimental studies within the previous 90 days prior to screening visit.
12. Patients having a pacemaker or other metal implants.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2026-03-01 (Estimated); Primary Completion 2027-03-01 (Estimated); Study Completion 2027-04-01 (Estimated)

PRIMARY OUTCOMES:
Change in Modified Fatigue Impact Scale (MFIS) total score | Baseline to End of Treatment (week 4)
  The Modified Fatigue Impact Scale (MFIS) is a 21-item patient-reported outcome assessing the impact of fatigue on physical, cognitive, and psychosocial functioning. Scores range from 0 to 84, with higher scores indicating greater fatigue impact. This outcome measures the change in MFIS total score from baseline to Week 4. Negative change values represent improvement in fatigue.

SECONDARY OUTCOMES:
Change in MFIS at Follow up | Baseline to Follow-up (week 8)
  MFIS is a 21-item patient-reported fatigue impact scale (range 0-84; higher scores indicate greater fatigue). This outcome assesses change in total MFIS score from baseline to follow-up assessment (Week 8).
Change in Fatigue Severity Scale (FSS) | Baseline to End of Treatment (week 4) and Follow-up (week 8)
  The Fatigue Severity Scale (FSS) is a 9-item questionnaire assessing the severity and functional impact of fatigue on daily activities. Each item is scored 1-7; the final score is the mean of all items, with higher scores indicating more severe fatigue. This outcome reflects change in FSS score from baseline to Week 4 and Week 8.
Change in Visual Analogue Scale for Mental Fatigue (VAS-MF) | Baseline to End of Treatment (week 4) and Follow-up (week 8)
  VAS-MF is a single-item 0-100 mm visual analogue scale measuring perceived mental fatigue. Higher values indicate greater fatigue. This outcome assesses change in VAS-MF score from baseline to Week 4 and Week 8
Change in PROMIS Fatigue Score | Baseline to End of Treatment (week 4) and Follow-up (week 8)
  The PROMIS Fatigue Short Form assesses self-reported fatigue and its interference with daily functioning. Scores are reported as standardized T-scores (mean 50, SD 10); higher scores indicate greater fatigue. This outcome measures change in PROMIS Fatigue from baseline to Week 4 and Week 8.
Change in Neuro-QoL Fatigue | Baseline to End of Treatment (week 4) and Follow-up (week 8)
  Neuro-QoL Fatigue evaluates the impact of fatigue on quality of life in neurological conditions. Scores are converted to T-scores (mean 50, SD 10), with higher scores indicating worse fatigue-related QoL. This outcome measures change in Neuro-QoL Fatigue from baseline to Week 4 and Week 8
Change in Symbol Digit Modalities Test (SDMT) | Baseline to End of Treatment (week 4) and Follow-up (week 8)
  The SDMT is a widely used measure of information processing speed. The score reflects the number of correct symbol-digit matches completed in 90 seconds, with higher scores indicating better cognitive performance. This outcome assesses change in SDMT score from baseline to Week 4 and Week 8.
Rate of Change in Daily Fatigue Severity (DFS) During the Treatment Period | Baseline through End of treatment (week 4)
  Daily Fatigue Severity (DFS) is assessed using a repeated self-reported rating of fatigue severity. Participants respond to the question "How fatigued do you feel today?" using a 7-point Likert scale, where higher scores indicate greater fatigue. This outcome assesses the rate of change in DFS across the treatment period to characterize longitudinal changes in daily fatigue.

OTHER OUTCOMES:
Change in MFIS Subscale Scores (Physical, Cognitive, Psychosocial) | Baseline to End of Treatment (week 4) and Follow-up (week 8)
  The MFIS yields three subscale scores assessing physical, cognitive, and psychosocial fatigue impact. Higher scores indicate greater impairment. This outcome measures change in each subscale from baseline to Week 4 and Week 8.
Cognitive Performance During Stimulation (Embedded Virtual Reality Tasks) | Baseline through End of Treatment (week 4)
  Cognitive performance is assessed using tasks embedded within the virtual reality environment during stimulation sessions. These tasks are designed to probe attention, processing speed, and learning dynamics while participants receive either active or sham stimulation. Performance data collected across sessions will be used for exploratory analyses of cognitive performance and learning trajectories during the treatment period.
Treatment Acceptability Ratings | Week 2, Week 4, and Week 8
  Longitudinal acceptability is evaluated at Weeks 2, 4 and 8 by asking participants about their willingness to use the device at home as a future treatment for MS-related fatigue. Responses provide insight into perceived usability, tolerability, and overall acceptability of the intervention over time.
Incidence of Adverse Events (AEs) | Baseline through Follow-up (week 8)
  AEs are defined as any unfavorable medical occurrence during the study, whether or not considered related to the intervention. Events are categorized by severity and relationship to study treatment. This outcome measures the proportion of participants experiencing at least one AE.
Incidence of Serious Adverse Events (SAEs) | Baseline through Week 8
  SAEs include events resulting in hospitalization, persistent disability, life-threatening conditions, or death. This outcome reports the number and proportion of participants experiencing SAEs during the study.
Tolerability: Session Attendance / Adherence Rate | Weeks 0-4
  Tolerability is assessed through adherence to the prescribed stimulation schedule. This outcome measures the percentage of completed sessions out of the total required (16 sessions delivered over 4 weeks).
Study Retention Rate | Baseline through Follow-up (week 8)
  Retention rate is defined as the proportion of participants who complete the follow-up assessment (week 8) relative to those enrolled.
Events of Clinical Interest (Agitation/Confusion) | Immediately monitored following stimulation; Through Week 4
  Events of clinical interest include agitation, confusion, or disorientation occurring within 1 hour of stimulation. This outcome captures their incidence and severity.

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital del Mar, Barcelona, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: No
This study collects pseudonymized clinical, behavioral, and EEG data that are subject to GDPR and local data protection regulations. Because the dataset contains sensitive information that cannot be fully de-identified, individual-level data will not be made publicly available. Aggregate results may be shared in publications or upon reasonable request to the sponsor.

REFERENCES:
- [Background] Reis C, Azizollahi H, Headley G, Navarro S, Hanslmayr S, Clouter A, Zanto TP, Certain R. VR-based gamma sensory stimulation: a pilot feasibility study. Sci Rep. 2025 Aug 5;15(1):28491. doi: 10.1038/s41598-025-13725-6. PMID 40764732
- [Background] Adaikkan C, Tsai LH. Gamma Entrainment: Impact on Neurocircuits, Glia, and Therapeutic Opportunities. Trends Neurosci. 2020 Jan;43(1):24-41. doi: 10.1016/j.tins.2019.11.001. Epub 2019 Dec 10. PMID 31836315
- [Background] Rodrigues-Amorim D, Bozzelli PL, Kim T, Liu L, Gibson O, Yang CY, Murdock MH, Galiana-Melendez F, Schatz B, Davison A, Islam MR, Shin Park D, Raju RM, Abdurrob F, Nelson AJ, Min Ren J, Yang V, Stokes MP, Tsai LH. Multisensory gamma stimulation mitigates the effects of demyelination induced by cuprizone in male mice. Nat Commun. 2024 Aug 8;15(1):6744. doi: 10.1038/s41467-024-51003-7. PMID 39112447